CLINICAL TRIAL: NCT02187679
Title: An Open Label, One Arm Pilot Study to Measure the Efficacy and Safety of Dysport in the Treatment of Vocal Tics in Patients With Tourette's Syndrome and Chronic Tic Disorders
Brief Title: Pilot Study for Use of Dysport in Treatment of Vocal Tics in Patients With Tourette's Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Detroit Clinical Research Center (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCRC-ISP0016888
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Tourette Syndrome; Chronic Vocal Tic
Keywords: Tourette Syndrome; Tourette's Syndrome; Chronic Vocal Tic; Vocal Tic
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — abobotulinumtoxinA

ARMS (1):
- Abobotulinum toxin A (Experimental): Abobotulinum toxin A Injection
  Interventions: Drug: Abobotulinum toxin A

INTERVENTIONS:
Drug: Abobotulinum toxin A
  Other Names: Dysport

SUMMARY:
Our intervention will be the injection of Abobotulinum toxin A into the affected site/vocal cords for patients with the diagnosis of Primary Tourette's syndrome. This is an efficacy trial to understand the right dosage of Abobotulinum toxin A which can be affective. The study will involve an injection of 2.5 units of Dysport on each side of the affected vocal cords for patients with a diagnosis of Primary Tourette's syndrome. The patients will also complete a self assessment survey on how vocal tics affect their daily lives. Afterward, a further evaluation of the tics will be conducted by the investigator using the Yale Global Tic Severity Scale. (YGTSS) evaluation. How this will be done is by a licensed ENT (Ear, Nose and Throat) physician. The windpipe will be number by a 2% lidocaine followed by a provoked cough by the patient. This will allow the lidocaine to be sprayed throughout the airway preventing coughing and swallowing during the procedure. An Electromyography (EMG) guidance a needle containing Dysport will be injected into the thyroarytenoid muscles will potentially reduce the vocal dyskinetic features in patients with TS. This needle will be connected to a syringe and once determined active, it will be placed appropriately when the EMG emits a characteristic sound. If this does not occur with the patient then the injection will be administered under direct vision via direct laryngoscopy using an orotracheal injector system.

This procedure is conducted in an outpatient clinic because no hospitalization is required. The patient is not allowed to consume food or drink for about 45-60 minutes after the injection. The throat will be numb and may cause coughing and some blood tinged sputum: The expectancy of this outcome is reason to not consider is a serious event. Asprin and ibuprofen is not allowed a week prior to and until the injection at least 3-4 days after to prevent excessive bleeding. The patient is also instructed to ensure that they chew their food thoroughly and drink sufficient water for the initial days after the study intervention. Mild dysphasia may be noted initially which should resolve within a few hours. On Visit 1, the patient will complete all required study documents and forms. Then the ENT physician will proceed with the injection Dysport on the same day. If unforeseen circumstances render the subject unable to be injected on the same day, the intervention must take place within three days and this will be considered V1, follow up events should be scheduled accordingly.

DETAILED DESCRIPTION:
The intervention for this pilot study will be the injection of Dysport (Abobotulinum toxin A) into the affected vocal cords for all patients with the diagnosis of Primary Tourette's syndrome. A total of 5 units of Dysport (on each side) will be administered to patients diagnosed with TS to determine whether they exhibit a reduction in the number of vocal tics. The patients will complete a self assessment survey about the manner in which the vocal tics are affecting their daily lives. Further evaluation of the tics will be conducted by the investigator using the Yale Global Tic Severity Scale (YGTSS) evaluation.

The intervention will be completed by a licensed ENT (Ears Nose and Throat) physician. The procedure will be conducted in an outpatient clinic setting because no hospitalization is required for this study. The windpipe will be numbed by a 2% lidocaine followed by a provoked cough by the patient. This will enable the lidocaine to be sprayed throughout the airway preventing any coughs or swallowing during the main intervention procedure. Under Electromyography (EMG) guidance a needle containing Dysport will be injected into the thyroarytenoid muscles which will potentially reduce the vocal dyskinetic features in individuals with TS. The needle containing Dysport will be connected to a syringe and once it is determined it is active, it will be placed appropriately when the EMG emits a characteristic sound. A total of 5 units of Dysport (2.5 units on each side) will be administered to the patient. If this does not occur with the patient then the injection will be administered under direct vision via direct laryngoscopy using an orotracheal injector system.

The patient will not be allowed to consume food or drink for approximately 45-60 minutes after Dysport has been injected. The throat will be numb after the anesthetic and may cause coughing and some blood tinged sputum which is expected and hence will not be considered a serious event. The patient will not be allowed to consume aspirin or ibuprofen a week prior to and till the intervention for at least 3-4 days after the intervention to prevent excessive bleeding. The patient will also be provided with specific instructions to ensure that they chew their food thoroughly and drink sufficient water for the initial days after the study intervention. Mild dysphasia may be noted initially which should resolve within a few hours.

On Visit 1 (Day 1), after the patient has completed all the required study documents and forms, the ENT physician will proceed with the injection of Dysport on the same day. However, if due to unforeseen circumstances, the subject cannot be injected on the same day, the intervention must take place within three days and this will be considered V1 (Day 1) and all follow up visits should be scheduled accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects between the ages of 18 and 65 with a primary clinical diagnosis of TS or chronic Tic Disorder with a duration of tics greater than one year.
* Subject is willing and able to provide informed consent. Subjects who are younger than age 21 must have written informed consent provided by the parent or legal guardian and assent provided by the patient when appropriate.
* Up to date tetanus immunization.
* Yale Global Tic Severity Scale score ≥20 with TS diagnosis or ≥14 for a Chronic Tic disorder.
* Female subjects of childbearing age must have a negative urine pregnancy test.

Exclusion Criteria:

* Patients who have a diagnosis of substance dependence disorder.
* Patients diagnosed with a significant and unstable major psychiatric disorder requiring treatment such as: Schizophrenia or Bipolar Disorder. Comorbid conditions such as: Obsessive Compulsive Disorder (OCD) and Attention Deficit Hyperactivity Disorder (ADHD) can be included.
* Patients diagnosed with the following types of Obsessive Compulsive Disorders: (All other types of obsessive compulsive disorders are acceptable)

  * Obsessive Compulsive Disorder for hand washing
  * Obsessive Compulsive Disorder for finger biting
  * Obsessive Compulsive Disorder for eye poking
  * Obsessive Compulsive Disorder for Dermatolomania
  * Obsessive Compulsive Disorder for Trichotillomania
  * Obsessive Compulsive Disorder for Head-Banging
* Patients with mental retardation.
* Patients diagnosed with progressive or degenerative neurological disorders or a structural disorder of the brain from birth, trauma or past infection.
* Patients taking more than one agent for the treatment of tics, more than one agent for the treatment of comorbid symptoms or more than one agent for the treatment of ADHD and/or the dose of the current treatment has not been stable for a minimum of 6 weeks.
* Female subjects who are pregnant or lactating.
* Allergy or hypersensitivity to Dysport or any other BoNT agent or their excipients
* Contraindications to treatment with any BoNT-A or BoNT-B preparations
* Based on Investigator opinion, patients in whom previous BoNT-A or BoNT-B therapy has failed to produce a clinical response or produced an intolerable adverse event
* Anticipated concomitant treatment with BoNT for other than TS
* Patients with sexually transmitted diseases such as: HIV, Herpes, Gonorrhea amongst others.
* Continuing Medications such as cholinergic medications.
* Autoimmune diseases like Myasthenia Gravis
* Unable or unwilling to maintain abstinence or use contraception for 28 days following all Dysport injections.
* Some forms of Cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Vocal Tic Reduction | 15 days
  Primary Outcome will be the reduction of tics as measured by the physician after 14 days and after 30 days. Only the Yale Global Tic Severity scale will be used to the measure the number of tics and their severity throughout the course of the study. These measurements will be compared with every visit to the score prior to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Dabrowski, MD, Principal Investigator — Detroit Clinical Research Center
Locations (1):
- Detroit Clinical Research Center, Farmington Hills, Michigan, United States